CLINICAL TRIAL: NCT05734079
Title: Impact of Digital Tools on the Quality of Bowel Preparation for Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Toni Ashqar, Dr. Toni Ashqar, Senior gastroenterologist, Ziv Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0085-22-ZIV
Record Dates: First submitted 2023-01-10; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Colonoscopy
Keywords: colonoscopy; gastroenterology; bowel preparation; digital; colorectal cancer screening
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (Active Comparator): Standard of care includes a written paper sheet that summarizes information about the colonoscopy procedure and bowel preparation.
  Interventions: Other: Standard of care
- Standard of care + Video call (Experimental): The video call will be performed at a designated time with a GE educated nurse. The purpose of the video call is (i) to clarify the patient in person about the colonoscopy procedure (ii) efficiently prepare the patient for bowel preparation by; asking the patient about her/his medical condition, the indication for colonoscopy, medical history, current medical status and medications currently taken. The patient will be inquired, whether she/he went through colonoscopy in the past, what preparation methods were undertaken and what the outcome of the examination was. Based on the information collected during the conversation, the designated nurse performing the interview will tailor the method of bowel preparation for the patient in terms of kind of relaxant, adjustment of medication intake and dietary adjustments before the examination.
  Interventions: Other: Standard of care + Video call
- Standard of care + Video call + Educational video film (Experimental): The video film will explain the colonoscopy procedure and the bowel preparation procedure, in layman's terms and in the patient's preferred language (Hebrew or Arabic).
  Interventions: Other: Standard of care + Video call + Educational video film

INTERVENTIONS:
Other: Standard of care — A written hand out containing all information required for bowel preparation
  Arms: Standard of care
Other: Standard of care + Video call — Standard of care and in addition a video call with a professional nurse conducted via digital devices and a free software (Zoom video communication or What's app application)
  Arms: Standard of care + Video call
Other: Standard of care + Video call + Educational video film — Standard of care and in addition to a video call, an explanatory short video on bowel preparation (video film), streamed to the patient's mobile device or computer
  Arms: Standard of care + Video call + Educational video film

SUMMARY:
This is a single blinded randomized controlled study. The main question of this study is whether better preparation by making full use of digital tools can increase patient compliance with the preparation methods for colonoscopy, and as a result improve bowel preparation quality and colonoscopy outcomes in a cost-effective manner.

Participants will randomly assigned to one of three colonoscopy preparation groups (i) a written hand out containing all information required for bowel preparation (standard care) (ii) standard care and in addition a video call with a professional nurse conducted via digital devices and a free software (Zoom video communication or What's app application) (iii) standard care and in addition to a video call as described above using an explanatory short video on bowel preparation (video film), streamed to the patient's mobile device or computer.

DETAILED DESCRIPTION:
Adequate bowel preparation is crucial for a successful and effective colonoscopy examination. Nevertheless, poor bowel preparation in patients is common and may lead to a lower quality of the examination that means a reduction in the rate of cecum intubation and lower detection rate of early and advanced adenoma. Finally, poor bowel preparation can lead to an abruption of the examination.

Digital advancement has been made in the context of colonoscopy bowel preparation, however high quality studies are still needed Ziv Medical Centre (ZMC) is a 300 bed governmental hospital located in Safed, Northern Israel that serves a diverse population. The gastroenterology department carries out approximately 1300 colonoscopies per year. A rapid audit has shown that approximately 15% of colonoscopies are stopped and up to 40% are incomplete, partly as a result of sub-optimal preparation.

The aim of this study is to determine whether better preparation by making full use of digital tools can increase patient compliance with the preparation methods for colonoscopy, and as a result improve bowel preparation quality and colonoscopy outcomes in a cost-effective manner.

This single blinded randomized controlled trial compares the effectiveness of bowel preparation in participants randomly assigned to one of three colonoscopy preparation groups (i) a written hand out containing all information required for bowel preparation (standard care) (ii) standard care and in addition a video call with a professional nurse conducted via digital devices and a free software (Zoom video communication or What's app application) (iii) standard care and in addition to a video call as described above using an explanatory short video on bowel preparation (video film), streamed to the patient's mobile device or computer.

All patients included in the trial will receive standard care 10 days before the examination. Patients randomized to the groups with a video call or a video call + video film will be contacted by a nurse to determine an appointment to the 10th day before examination. Patients randomized to the study arm including an educational video film will be sent a link to the video film after the video call. On the day of the exam, during the examination, the medical doctor records an OBPS score as described. After the exam, the medical doctor will register whether the exam was complete, incomplete, stopped and whether hospitalization was needed. After the examination and recovery, all patients will receive a short satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* access to a digital device (smart phone, tablet, personal computer, laptop- this includes individuals who can use devices from household of relatives)
* ability to understand instructions in Hebrew or Arabic
* ability to sign a digital consent

Exclusion Criteria:

• pregnancy (first trimester)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 825 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The Ottawa Bowel Preparation Scale (OBPS) | OBPS will be evaluated during the colonoscopy procedure
  A standard method used to assess a patient's bowel preparation for colonoscopies. The bowel preparation score is a sum of a segmental score (right-colon, mid-colon and rectosigmoid-colon) and a fluid quantity score. The segmental score is quantified on a scale of 0 to 4, with; 0 indicating perfect cleansing, 1 indicating good cleansing, 2 indicating Fair cleansing, 3 indicating poor cleansing and 4 indicating inadequate cleansing. Overall fluid quantity is quantified on a scale of 0 to 2, with; 0 indicating no fluid in the colon and 2 indicating a large amount of fluid in the colon. Both the colon score and fluid score result in an overall score ranging from 0 to 14, with; 0 an Excellent cleansing quality and 14 indicates the worst cleansing quality. Estimations of the scores are made by the medical doctors during the exam and are fed into a commercial software that calculates the overall OBPS score.

SECONDARY OUTCOMES:
Patient's satisfaction questionaire | Questionnaires will be given to the patients immediately after the colonoscopy
  Patients will be asked about various aspects of the preparation using likert scales- the scores for each question will be compared across groups. The questionaires will include several questions about demographic background such as education level and occupation.
Colonoscopy completion | Colonoscopy completion will be recorded for 1 year
  The proportion of successfully completed colonoscopies will be quantified.
The proportional change in the annual cost of treatment services | 1 year
  The proportional change in the annual cost of running the service will be calculated, taking into account costs (research nurse, cost of developing the video etc.) and saving (averted complications, failed colonoscopies requiring re-booking etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Ashqar, Dr., Principal Investigator — Ziv Medical Center

IPD SHARING:
Plan to Share IPD: No